CLINICAL TRIAL: NCT03882411
Title: An Information tecHnology Approach to implEmenting Depression treAtment in caRdiac patienTs: [iHeartDepCare Trial]
Brief Title: An IT Approach to Implementing Depression Treatment in Cardiac Patients (iHeart DepCare)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nathalie Moise, Assistant Professor of Medicine, Dept of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAR9175 - III; 1R01HL141609-01 (NIH)
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms; Coronary Heart Disease
Keywords: Implementation science
MeSH Terms: conditions — Depression; Coronary Disease | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Pre-post single group design with 8 clinic clusters randomized to timing of receipt of intervention with patients nested within providers nested within clinic clusters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electronic shared decision making (eSDM) Tool (Experimental): In the pre-intervention period, patients in clinic clusters will receive usual care.
  When a clinic cluster's randomly allotted intervention period arrives, coronary heart disease patients in that given clinic cluster will complete a web application, which delivers screening, behavioral activation and shared decision making (eSDM), and providers will receive education and a patient preference report generated from the application.
  During both the pre and post intervention periods, patients will be assessed at baseline and 6 month follow up.
  Interventions: Behavioral: Electronic shared decision making (eSDM) tool

INTERVENTIONS:
Behavioral: Electronic shared decision making (eSDM) tool — The web application includes depression screening, behavioral activation, and a patient preference driven treatment selection decision aid. Treatment options will include medications, cardiac rehab/exercise program, and therapy. In addition to education, providers will receive a patient preference report in real time with options for coordination of care
  Other Names: eSDM intervention

SUMMARY:
The purpose of this study is to examine the effect of a brief electronic shared decision making (eSDM) intervention on depressive symptoms in coronary heart disease patients with elevated depressive symptoms.

DETAILED DESCRIPTION:
Depression is common in patients with coronary heart disease and associated with increased cardiac morbidity and mortality. Treating depressive symptoms appears to improve depressive symptoms and quality of life. Despite expert recommendations to screen and treat depressive symptoms fewer coronary heart disease patients engage in depression treatment than the general population, perhaps due to 1) sub-optimal provider awareness and referral rates and 2) low self-efficacy, stigma and misattribution of depressive symptoms among coronary heart disease patients. In addition, few real world theory-informed implementation trials exist for improving screening and treatment in outpatient settings.

The specific aim is to determine whether an electronic shared decision making (eSDM) and behavioral activation tool improves depressive symptoms and treatment initiation in coronary heart disease patients with elevated depressive symptoms. To accomplish these aims, a hybrid effectiveness-implementation trial will be conducted using a pre-post design across socioeconomically diverse cardiology and primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary heart disease
* English or Spanish Speaking
* Elevated Depressive symptoms (PHQ9 ≥10)
* Appointment at participating cardiology or primary care clinics

Exclusion Criteria:

* Under the care of a psychiatrist [**On 6/22/2022, this exclusion criteria was removed for those clusters of clinics not already in the post-implementation period**]
* Diagnosis/history of psychosis or schizophrenia
* Diagnosis/history of bipolar disorder
* Attempted suicide
* Non-English or Spanish speaking
* Dementia or severe cognitive impairment
* Non-elevated depressive symptoms
* Alcohol or substance abuse
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Beck Depression Index (BDI-II) | Baseline, Follow-up visit (approximately 6 months)
  Change in total BDI (21-item measure of depressive symptoms [0-63]; higher score constitutes worse burden of symptoms) from baseline to follow visit during the pre-intervention period compared to post-intervention period

SECONDARY OUTCOMES:
Proportion of patients who initiate treatment | Baseline, Follow-up visit (approximately 6 months)
  Proportion of enrolled patients who initiate any depression treatment (medications, cardiac rehab/exercise program, therapy) from baseline to follow up visit in the pre-intervention compared to post-intervention period
Mean Patient Activation | Baseline
  Mean baseline patient activation measure [PAM] (13-items, range 0-100, higher score indicates greater activation] in the pre-intervention compared to post-intervention period
Mean Decisional Conflict Scale | Baseline
  Mean decisional conflict (measures personal perceptions of uncertainty around choosing among treatment option, 10 items, range 0-100, higher score indicates greater conflict) of patients.
Mean change in quality of life (QoL) | Baseline, Follow-up visit (approximately 6 months)
  Change in QoL from from baseline to follow up visit in the pre-intervention compared to post-intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Moise, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No